CLINICAL TRIAL: NCT06281340
Title: Changes in Intra-articular Parameters by Doppler Ultrasound in Patients With Hemophilic Ankle Arthropathy After Manual Therapy Intervention: A Randomized Double-blind Clinical Study
Brief Title: Changes in Intra-articular Parameters by Doppler Ultrasound in Patients With Hemophilic Ankle Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: He-ankle US
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Hemophilia
Keywords: Hemophilia; Ankle; Manual therapy; Ultrasound; Joint pain; Joint damage
MeSH Terms: conditions — Hemophilia A; Arthralgia | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Randomization will be performed using a computerized randomization procedure by permuted blocks of 4 subjects in each recruitment center. The 6 possible sequence alternatives will be modified in each block. This task will be carried out by a person who is not involved in the study and who will not know the identity of the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patients included in the experimental group will receive a session of manual physiotherapy using joint gliding techniques, myofascial and manipulative techniques of the tobioperoneoastotalar and subtalar joints. The intervention will be performed on both ankles.
  Interventions: Other: Manual therapy
- Control group (Placebo Comparator): Patients included in the control group will receive a placebo manual physical therapy session, simulating joint sliding techniques, myofascial and manipulative techniques of the tobioperoneoastotalar and subtalar joints, without any stimulus other than the pressure exerted by the physical therapist with his hands when mobilizing the foot. The placebo intervention will be performed on both ankles.
  Interventions: Other: Placebo manual therapy

INTERVENTIONS:
Other: Manual therapy — Each session will last approximately 50-60 minutes. Each session is composed of 10 techniques, 9 of which correspond to manual interventions commonly used in the field of manual therapy and adapted to patients with hemophilic arthropathy, according to the criteria previously established in studies that assess the safety of manual interventions in hemophilic arthropathy.
  Arms: Experimental group
Other: Placebo manual therapy — Each session will last approximately 50-60 minutes. Each session consists of the placebo application of 10 techniques, 9 of which correspond to manual interventions commonly used in the field of manual therapy and adapted to patients with hemophilic arthropathy, according to criteria previously established in studies that assess the safety of manual interventions in hemophilic arthropathy. In the techniques there will be no joint sliding, manipulations or myofascial inductions, being the only stimulus the contact of the physiotherapist with his hands and the pressure exerted with these, on the ankle.
  Arms: Control group

SUMMARY:
Introduction: Hemophilic ankle arthropathy is manifested by functional degenerative alterations, intra-articular alterations, and chronic pain. Manual therapy techniques are used in the treatment of hemophilic ankle arthropathy for the improvement of pain and mobility.

Design. Double-blind randomized pilot trial. Aimed: To evaluate the ultrasound changes by means of Doppler imaging after manual therapy intervention.

Patients: A total of 20 adult patients with hemophilic ankle arthropathy will be recruited.

Intervention: Each manual therapy session will last approximately 50 minutes, with 1 session per week for a period of 3 weeks. The treatment program includes 10 techniques that will be administered bilaterally.

Measuring instruments: Patients will be evaluated qualitatively with ultrasound (HEAD-US scale) and assessment with Doppler ultrasound. The clinical variables will be joint damage (Hemophilia Joint Health Score) and pain intensity (Visual Analogue Scale).

Expected results: Check the safety of manual therapy in patients with hemophilia regarding subclinical bleeding. Assess changes related to joint inflammatory state with imaging techniques. Observe changes in pain intensity and joint damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A or B.
* Persons over 18 years of age.
* Patients with a medical diagnosis of ankle arthropathy (with clinical assessment of more than 4 points on the Hemophilia Joint Health Score.
* Patients on prophylactic or on-demand treatment with FVIII / FIX concentrates.
* Sign the informed consent document.

Exclusion Criteria:

* Patients with inhibitors (antibodies against FVIII or FIX) without treatment with monoclonal antibodies.
* Patients with neurological or cognitive alterations that impede the comprehension of questionnaires and physical tests.
* Patients who have developed an ankle hemarthrosis in the 3 months prior to the study.
* Patients who at the time of the study are receiving ankle physiotherapy treatment.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline sonographic changes after 4 hours | Screening visit and after four hours follow-up
  Ultrasound changes will be measured with the Haemophilia Early Arthropathy Detection with UltraSound score. This scale evaluates two parameters: i) inflammatory activity (scores synovial hypertrophy from 0 to 2 points depending on whether involvement is identified); and ii) involvement of articular surfaces (assesses articular cartilage and bone involvement). In the assessment of articular cartilage, a score from 0 to 4 is established (0: normal; 4: complete destruction of cartilage or cannot be visualized). Bone is scored from 0 to 2 points (0: normal; 2: involvement with osteophytes).

SECONDARY OUTCOMES:
Change from baseline joint pain after 4 hours | Screening visit and after four hours follow-up
  The intensity of ankle joint pain will be measured with the visual analog scale. This scale has shown moderate reliability (ICC: 0.60-0.77) in patients with chronic musculoskeletal pain. Its scores range from 0 to 10 points (from no pain to the maximum pain perceived by the patient).
Change from baseline joint damage after 4 hours | Screening visit and after four hours follow-up
  Joint damage will be measured with the Hemophilia Joint Health Score (HJHS). This measurement instrument will be used to assess the joint status of both ankles. It includes 8 items (swelling and duration of swelling, pain, muscle atrophy and strength, crepitus, and loss of flexion and extension) with a range of 0 to 20 points per joint (the higher the score, the greater the joint impairment).
Change from baseline degree of joint inflammation after 4 hours | Screening visit and after four hours follow-up
  With a doppler assessment, a qualitative assessment of the degree of joint inflammation (semi-quantitative visual scale from 1 to 4: none, mild, moderate, severe) and a quantitative assessment by quantifying the resistance index (RI) will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain